CLINICAL TRIAL: NCT05786040
Title: Phase II Study to Assess the Efficacy of Combined Tafasitamab and Rituximab in Front-Line Treatment of Post-Transplant Lymphoproliferative Disorder
Brief Title: Tafasitamab and Rituximab for Front-Line Treatment of Post-Transplant Lymphoproliferative Disorder
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Timothy Voorhees (Other)
Responsible Party: Sponsor-Investigator, Timothy Voorhees, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-22114; NCI-2023-02048 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2023-03-13; First posted 2023-03-27 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Monomorphic B-Cell Post-Transplant Lymphoproliferative Disorder; Polymorphic Post-Transplant Lymphoproliferative Disorder
MeSH Terms: interventions — Biopsy; Specimen Handling; Magnetic Resonance Spectroscopy; Rituximab; CT-P10; tafasitamab; Immunoglobulins; Disulfides

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (tafasitamab, rituximab) (Experimental): Patients receive tafasitamab IV and rituximab IV or SC on study. Patients who have CR or PR after 4 cycles may receive additional tafasitamab and rituximab on study. Patients also undergo PET or CT, biopsy, and collection of blood samples throughout the trial.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Positron Emission Tomography; Biological: Rituximab; Biological: Tafasitamab

INTERVENTIONS:
Procedure: Biopsy — Undergo biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Procedure: Positron Emission Tomography — Undergo PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Biological: Rituximab — Given IV or SC
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Riabni; Rituxan; Rituximab ABBS; Rituximab ARRX; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; Rituximab Biosimilar SIBP-02; rituximab biosimilar TQB2303; Rituximab PVVR; rituximab-abbs; Rituximab-arrx; Rituximab-pvvr; RTXM83; Ruxience; Truxima
Biological: Tafasitamab — Given IV
  Other Names: Immunoglobulin, Anti-(Human Cd19 Antigen) (Human-mus musculus Monoclonal MOR00208 Heavy Chain), Disulfide with Human-mus musculus Monoclonal MOR00208 .Kappa.-chain, Dimer; Monjuvi; MOR-00208; MOR00208; MOR208; Tafasitamab-cxix; XmAb5574

SUMMARY:
This phase II trial tests how well tafasitamab and rituximab work for front-line treatment of patients with post-transplant lymphoproliferative disorder. Post-transplant lymphoproliferative disorder (PTLD) is the name for types of lymphoma that sometimes develop in people who have had a transplant. It can affect people who are taking medicines to suppress their immune system. Tafasitamab injection is in a class of medications called monoclonal antibodies. It works by helping the body to slow or stop the growth of cancer cells. Rituximab is a monoclonal antibody. It binds to a protein called CD20, which is found on B cells (a type of white blood cell) and some types of cancer cells. This may help the immune system kill cancer cells. Giving the combination of tafasitamab and rituximab may work better in treating patients with post-transplant lymphoproliferative disorder.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To estimate the rate of complete response (CR) after 4 cycles of weekly (or 7-day) treatments with combined rituximab and tafasitamab in subjects with post-transplant lymphoproliferative disorder (PTLD).

SECONDARY OBJECTIVES:

I. To describe the safety profile of treatment with combined rituximab and tafasitamab in subjects with PTLD.

II. To estimate the objective response rate (ORR), defined as clinical response (CR + partial response [PR]) after 4 cycles of weekly (or 7-day) treatments with combined rituximab and tafasitamab in subjects with PTLD.

III. To determine the best overall response (BOR), defined as best clinical response (CR + PR) at either the completion of 4 cycles of weekly (or 7-day) treatments or 4 consolidation cycles (every 3 week) of combined rituximab and tafasitamab in subjects with PTLD.

IV. To estimate the rate of complete response (CR) after completion of consolidation treatments of combined rituximab and tafasitamab in subjects with PTLD.

V. To estimate the progression free survival (PFS) in subjects with PTLD treated with rituximab and tafasitamab.

VI. To estimate the overall survival (OS) in subjects with PTLD treated with rituximab and tafasitamab.

EXPLORATORY OBJECTIVES:

I. To describe baseline CD19 and CD20 expression on malignant lymphocytes by flow cytometry in subjects with PTLD.

II. To describe the relationship of tumor microenvironment characteristics using ribonucleic acid sequencing (RNASeq) with clinical response to combined rituximab and tafasitamab in subjects with PTLD.

III. To characterize the peripheral immunophenotype changes using cytometry by time-of-flight (CyTOF) from cycle 1 (C1) day 1 (D1) to cycle 5 (C5)D1 of combined rituximab and tafasitamab in subjects with PTLD.

IV. To describe the type of immunosuppression and amount reduced in subjects with PTLD.

V. To describe the relationship between metabolic tumor volume at diagnosis and response to combined rituximab and tafasitamab in subjects with PTLD.

VI. To characterize Epstein-barr virus (EBV) methylation alterations in EBV positive PTLDs.

OUTLINE:

Patients receive tafasitamab intravenously (IV) and rituximab IV or subcutaneously (SC) on study. Patients who have CR or PR after 4 cycles may receive additional tafasitamab and rituximab on study. Patients also undergo positron emission tomography (PET) or computed tomography (CT), biopsy, and collection of blood samples throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained to participate in the study and Health Insurance Portability and Accountability Act (HIPAA) authorization for release of personal health information
* Age >= 18 years at the time of consent
* Karnofsky scale > 30% or Eastern Cooperative Oncology Group (ECOG) =< 3 (can be assessed after pre-phase steroids)
* Histological evidence of B-cell PTLD (monomorphic and polymorphic) following solid organ transplantation; expresses CD19 and CD20, with or without EBV association, confirmed after biopsy or resection of tumor
* Measurable disease of > 1.5 cm in diameter and/or bone marrow involvement
* Subjects having undergone heart, lung, liver, kidney, pancreas, small intestine transplantation or a combination of the organ transplantations mentioned
* No prior lines of therapy for PTLD (palliative radiation, steroids, antiviral therapy, and reduction in immunosuppression are allowed)
* Human immunodeficiency virus (HIV) infection is allowed if viral load is undetectable at time of enrollment and CD4+ count > 200 cells/uL
* Expected survival greater than 30 days
* Absolute neutrophil count (ANC) >= 1.0 x 10^9/L (obtained within 14 days prior to initiating study treatment)

  * Note: Hematology and other lab parameters that are =< grade 2 BUT still meet criteria for study entry are allowed. Furthermore, changes in laboratory parameters during the study should not be considered adverse events unless they meet criteria for dose modification(s) of study medication outlined by the protocol and/or worsen from baseline during therapy
* Platelets >= 50 x 10^9/L (obtained within 14 days prior to initiating study treatment)

  * Note: Hematology and other lab parameters that are =< grade 2 BUT still meet criteria for study entry are allowed. Furthermore, changes in laboratory parameters during the study should not be considered adverse events unless they meet criteria for dose modification(s) of study medication outlined by the protocol and/or worsen from baseline during therapy
* Creatinine clearance (mL/min) >= 30 mL/min (obtained within 14 days prior to initiating study treatment)

  * Cockcroft-Gault Equation
  * Note: Hematology and other lab parameters that are =< grade 2 BUT still meet criteria for study entry are allowed. Furthermore, changes in laboratory parameters during the study should not be considered adverse events unless they meet criteria for dose modification(s) of study medication outlined by the protocol and/or worsen from baseline during therapy
* Bilirubin =< 3.0 x upper limit of normal (ULN). Subjects with Gilbert's syndrome may be enrolled despite a total bilirubin level > 3.0 mg/dL if their conjugated bilirubin is =< 3.0 x ULN) (obtained within 14 days prior to initiating study treatment)

  * Note: Hematology and other lab parameters that are =< grade 2 BUT still meet criteria for study entry are allowed. Furthermore, changes in laboratory parameters during the study should not be considered adverse events unless they meet criteria for dose modification(s) of study medication outlined by the protocol and/or worsen from baseline during therapy
* Aspartate aminotransferase (AST) =< 3.0 x ULN (obtained within 14 days prior to initiating study treatment)

  * Note: Hematology and other lab parameters that are =< grade 2 BUT still meet criteria for study entry are allowed. Furthermore, changes in laboratory parameters during the study should not be considered adverse events unless they meet criteria for dose modification(s) of study medication outlined by the protocol and/or worsen from baseline during therapy
* Alanine aminotransferase (ALT) =< 3.0 x ULN (obtained within 14 days prior to initiating study treatment)

  * Note: Hematology and other lab parameters that are =< grade 2 BUT still meet criteria for study entry are allowed. Furthermore, changes in laboratory parameters during the study should not be considered adverse events unless they meet criteria for dose modification(s) of study medication outlined by the protocol and/or worsen from baseline during therapy
* Females of childbearing potential must have a negative serum pregnancy test within 3 days prior to registration. NOTE: Females are considered of childbearing potential unless they are surgically sterile (have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are naturally postmenopausal for at least 12 consecutive months. Documentation of postmenopausal status must be provided
* Females of childbearing potential must be willing to abstain from heterosexual activity or to use 2 forms of effective methods of contraception from the time of informed consent until 12 months after treatment the last dose of rituximab or tafasitamab. The two contraception methods can be comprised of two barrier methods, or a barrier method plus a hormonal method or an intrauterine device that meets < 1% failure rate for protection from pregnancy in the product label
* Male subjects with female partners must have had a prior vasectomy or agree to use an adequate method of contraception (i.e., double barrier method: condom plus spermicidal agent) starting with the first dose of study therapy through 12 months after the last dose of rituximab
* Subjects with prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the experimental regimen are eligible for the trial
* Subject is willing and able to comply with study procedures based on the judgement of the investigator or protocol designee

Exclusion Criteria:

* Uncontrolled active infection. Patients requiring systemic therapy are eligible if the infection is deemed controlled by the investigator
* Post-transplant lymphoproliferative disorder following liquid transplantation
* Pregnant or breastfeeding (NOTE: breast milk cannot be stored for future use while the mother is being treated on study and lactating females must agree to not breastfeed while taking study drugs)
* Subjects with central nervous system (CNS) involvement by PTLD
* Uncontrolled concomitant illness including, but not limited to, symptomatic congestive heart failure (New York Heart Association [NYHA] class III or IV), unstable angina pectoris, myocardial infarction within 1 month prior to enrollment, uncontrolled cardiac arrhythmias, uncontrolled seizures, or severe non-compensated hypertension (systolic blood pressure >= 180 mmHg or diastolic blood pressure >= 120 mmHg)
* History of progressive multifocal leukoencephalopathy
* Active hepatitis B infection with positive viral polymerase chain reaction (PCR) from the blood. Subjects with active hepatitis B infection and undetectable viral PCR from the blood will be allowed with concurrent use of entecavir suppression
* Prior treatment for PTLD with the exception of radiation, antivirals, steroids and reduced immunosuppression
* Electrocardiogram (ECG) abnormality at screening has to be documented by the investigator as not medically relevant
* Any condition, including the presence of laboratory values which is deemed by the clinician to place the subject at an unacceptable risk or confounds the ability to interpret the data from this study
* Live virus vaccines must not be administered within 28 days of the start of study treatment
* Any investigational treatments must have been completed at least 7 days prior to the start of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-03-23 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of patients who achieve a complete response (CR) | within 1 week after 4 cycles of combined therapy
  Assessed using Lugano criteria. Will be calculated as the number of patients who achieve CR divided by the number of evaluable patients, and presented with the 95% binomial confidence interval.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 28 days after the last dose of tafasitamab and rituximab
  Adverse events will be described and classified per the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 guidelines. The maximum grade of each type of toxicity will be extracted for each patient, and frequency counts will be tabulated to determine toxicity patterns, especially for grade 3 or above adverse events.
Overall response rate | Up to 3 years
  Defined as clinical response (CR + partial response [PR]) after 4 cycles of weekly (or 7-day) treatments with combined rituximab and tafasitamab using Lugano criteria.
Best overall response | Up to 3 years
  Defined as best clinical response (CR + PR) at the completion of either 4 cycles of weekly (or 7-day) treatments or 4 consolidation cycles (every 3 week) of combined rituximab and tafasitamab using Lugano criteria. Will be estimated and 95% confidence interval computed.
Rate of CR after completion of consolidation treatments | Up to 3 years
  Will be estimated and 95% confidence interval computed.
Progression free survival | From the date of treatment initiation to date of progression or death, whichever occurs first, censoring patients who are alive without progression at time of last known follow-up, assessed up to 3 years
  Will be estimated using the Kaplan-Meier method.
Overall survival | From date of treatment initiation to date of death due to all causes, and censoring alive patients at date of last known follow-up, assessed up to 3 years
  Will be estimated using the Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy J Voorhees, MD, MSCR, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (3):
- United States (3):
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - University of North Carolina-Hillsborough Campus, Hillsborough, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu